CLINICAL TRIAL: NCT01613703
Title: Open-Label, Single-Center, Single Dose Positron Emission Topography (PET) Using [11C]PBR28 to Evaluate Brain Translocator Protein 18KDa (TSPO) Occupancy of ONO-2952 in Healthy Adult Subjects
Brief Title: ONO-2952 Single-dose PET Study in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-2952POU003
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-2952; Healthy adult subjects; single doe; PET study; Safety; Tolerability
MeSH Terms: interventions — ONO-2952

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: ONO-2952

INTERVENTIONS:
Drug: ONO-2952 — 1 mg to 200 mg QD at a single descending dose

SUMMARY:
The primary objective of this study is to evaluate the brain TSPO occupancy of ONO-2952 in healthy adult subjects after a single dose using [11C]PBR28 as a specific PET ligand for TSPO. The secondary objective is to evaluate the relationship between TSPO occupancy and the plasma concentration of ONO-2952 and to investigate the safety and tolerability of ONO-2952 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male or female subjects (18-55 inclusive)
* Body mass index (BMI) of 19-35 kg/m2 (inclusive)
* For females, surgically sterilized, postmenopausal, or who are non- lactating and agree to use a double barrier method of contraception

Exclusion Criteria:

* History or presence of clinically significant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the brain TSPO occupancy of ONO-2952 in healthy adult subjects after a single dose using [11C]PBR28 as a specific PET ligand for TSPO | 2 days

SECONDARY OUTCOMES:
To evaluate the relationship between TSPO occupancy and the plasma concentration of ONO-2952 | 2 days
To investigate the safety and tolerability of ONO-2952 in healthy adult subjects | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Pittsburgh Clinical Site, Pittsburgh, Pennsylvania, United States